CLINICAL TRIAL: NCT03867799
Title: Immunotherapy Sequencing in COlon and REctal Cancer
Brief Title: iSCORE: Immunotherapy Sequencing in COlon and REctal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4938
Record Dates: First submitted 2019-01-30; First posted 2019-03-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Relatlimab (Experimental): Nivolumab 480mg and Relatlimab 160mg will be administered intravenously every 4 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Immunotherapy
  Other Names: Relatlimab

SUMMARY:
This is a single-arm, single centre open-label, phase II interventional clinical trial of combination immunotherapy with Nivolumab and Relatlimab in mCRC.

DETAILED DESCRIPTION:
This is a single-arm, single centre open-label, phase II interventional clinical trial of combination immunotherapy with Nivolumab and Relatlimab in mCRC.

Patients with metastatic RAS/RAF WT colorectal cancer who have previously had a radiological response to EGFR inhibitors i.e. Cetuximab or Panitumumab, either combined with chemotherapy or as single agents, but subsequently experienced progression of their disease will be eligible for the study. They will consent to the study ideally within 3 months having progressed/ become refractory to EGFR blockable and undergo a mandatory baseline biopsy within this time period.

Patients will receive Nivolumab and Relatlimab every 4 weeks and will start on study treatment as soon as possible after the baseline biopsy. After starting on the study drugs, there will be a mandatory 'on-treatment' biopsy at day 21 ± 3 days. Response assessments in the form of either CT or MRI scans will take place every 8 weeks throughout the study for the 12 months and every 12 weeks from 12 months onwards. Patients will continue on the study until progressive disease (PD) is confirmed by RECIST 1.1 or when maximum duration of treatment of 24 months has been reached

There will be the possibility of 'treating beyond progression' if participants are deriving clinical benefit from treatment to encompass the possibility of pseudoprogression. At PD participants will undergo a further biopsy. The investigators envisage enrolling a total of 25 participants and the investigators anticipate 30 months as a feasible time frame for accrual.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients aged ≥18 years
2. Patients with histologically confirmed advanced/metastatic RAS/RAF wild type colon or rectal adenocarcinoma who had a prior radiological response to EGFR blockade as a single agent or in combination with chemotherapy but have subsequently progressed/ become refractory to this treatment based on physician judgment. Patients should not have received any other systemic anti-cancer therapy between the end of treatment with EGFR inhibitors as a single agents or in combination with chemotherapy and screening for the iSCORE study
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Estimated life expectancy of at least 3 months at the time of informed consent per Investigator assessment
5. Adequate organ functioning as defined by the following:

   i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (stable off any growth factor within 4 weeks prior to first study drug administration) ii. Platelet count ≥ 100 × 109/L (Transfusion to achieve this level is not permitted within 2 weeks of first study drug administration) iii. Haemoglobin ≥ 8.5 g/dL (Transfusion to achieve this level is not permitted within 2 weeks of first study drug administration) iv. Creatinine < 1.5 X ULN or creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula) v. AST and ALT levels ≤ 3 × ULN vi. Lipase and amylase < 1.5 ULN vii. Total bilirubin level ≤ 1.5 ULN (except patients with Gilbert's Syndrome who must have a normal direct bilirubin) viii. Normal thyroid function or on stable hormone supplementation per investigator assessment ix. Albumin >28 g/dL x. LVEF assessment with documented LVEF ≥ 50% by TTE within 6 months from first study drug administration
6. Negative serum or urine pregnancy test at screening for women of childbearing potential**
7. Highly effective contraception for both male and female patients throughout the study and for at least 165 days for women 225 days for males after the last treatment administration if the risk of conception exists. Please refer to Section 9.15 - Pregnancy reporting for details of acceptable and unacceptable methods of contraception.
8. Patient must consent and be eligible to undergo mandatory baseline and sequential biopsies; in such case as a specimen cannot be obtained at acceptable clinical risk as judged by the Investigator then patients may still be included in the study. Patients must not be anti-coagulated at the time of biopsy or on aspirin/clopidogrel for 7 days pre-biopsy
9. Resolved acute effects of prior therapy to baseline severity or ≤Grade 1 except for AEs not constituting a safety risk by investigator judgement
10. Signed and dated informed consent
11. Patients willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other procedures. Prisoners and patients who are involuntarily incarcerated are excluded
12. Presence of measurable disease as defined by RECIST v 1.1 criteria for response assessment ** Defined as a pre-menopausal female capable of becoming pregnant. This includes women on oral, injectable or mechanical contraception

Exclusion Criteria

Patients are not eligible for the trial if any of the exclusion criteria below are met:

1. Systemic therapy within 4 weeks prior to the planned administration of the first study treatment dose
2. Major surgery within 4 weeks or radiation therapy within 14 days prior to study entry. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed 48 hours prior to study entry and there is at least one measurable lesion that has not been irradiated
3. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation
4. Previous exposure to immune checkpoint inhibitors or immune co-stimulatory drugs such as but not limited to anti-CTLA-4, anti-PD-1, anti-PDL1, anti-PD-2, anti-KIR, anti-CD137, anti-LAG-3, anti-OX40 antibodies or IDO or CXCR2 targeted agents
5. Known severe hypersensitivity reactions (Grade ≥ 3 NCI CTCAE v 5.0) to monoclonal antibodies or related compounds or any of their components (e.g. history of severe hypersensitivity reactions to drugs formulated with polysorbate 80), any history of anaphylaxis or uncontrolled asthma (defined a 3 or more features of partially controlled asthma)
6. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
7. Active infection requiring systemic therapy
8. Any active malignancy, with the exception of adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer or other locally curable cancers including superficial bladder cancer, carcinoma in situ of the prostate, cervix or breast
9. Significant acute or chronic infections including, among others:

   * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
   * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
10. All patients with brain metastases, except those meeting the following criteria:

    * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrolment
    * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
    * Patients must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)
11. Prior organ transplantation, including allogeneic stem cell transplantation
12. Any active autoimmune disease that has required systemic treatment in past 2 years (i.e, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
13. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

    1. Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
    2. Uncontrolled angina within the 3 months prior to consent
    3. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes, or poorly controlled atrial fibrillation)
    4. QTc prolongation > 480 msec
    5. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc )
    6. Cardiovascular disease-related requirement for daily supplemental oxygen
    7. History of two or more MIs OR two or more coronary revascularization procedures
    8. Patients with history of myocarditis, regardless of aetiology
14. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Patients with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 x ULN. If TnT or TnI levels are >1 to 2 × ULN within 24 hours, the patient may undergo a cardiac evaluation and be considered for treatment based on the discretion of the PI. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the patient may undergo a cardiac evaluation and be considered for treatment, based on the discretion of the CI
15. Patients with a history of interstitial lung disease or radiological evidence of pulmonary fibrosis
16. Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1) except alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
17. Pregnancy or lactation (females of childbearing potential must have a negative pregnancy test within 3 days prior to treatment initiation and every month during treatment
18. Known alcohol or drug abuse
19. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
20. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
21. Vaccination within 4 weeks of the first dose of study drugs and while on trial is prohibited except for administration of inactivated vaccines
22. A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 6 months from treatment initiation

SECONDARY OUTCOMES:
NCI CTCAE version 5.0 toxicity | within 30 days of the last dose of study treatment
Disease Control Rate (DCR) | 12 and 24 months
Duration of disease control | 6, 12 and 24 months
Best Objective Response Rate | 6, 12 and 24 months
Progression Free Survival | Time from registration to progression (radiological or clinical) or death at 6 months, 12 months and 24 months
Overall survival | time from registration to death from any cause at 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No